CLINICAL TRIAL: NCT01552785
Title: A Comparison of Measurements of Peripheral Tissue Oxygenation by NONIN EQUANOX 7600, INVOS 5100c, and FORE-SIGHT
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gorm Greisen, Professor, Rigshospitalet, Denmark
Other Study IDs: NIF010312
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Near Infrared Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adults
  Interventions: Device: Peripheral near infrared spectroscopy

INTERVENTIONS:
Device: Peripheral near infrared spectroscopy — Devices: NONIN 7600 EQUANOX with sensor Model 8004CA, INVOS 5100c with SAFB-SM, and FORE-SIGHT with medium sensor

SUMMARY:
A comparison of three different devices using near infrared spectroscopy to measure the regional oxygenation. Both absolute values, reproducibility of measurements and sensitivity to changes will be estimated. The study hypothesis is that NONIN EQUANOX 7600 with sensor Model 8004CA, INVOS 5100c with sensor SAFB-SM and FORE-SIGHT with medium sensor have similar characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Double skin fold less than 1 cm on the lower arm

Exclusion Criteria:

* Chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Citizens of Copenhagen
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Absolute mean value of peripheral regional tissue oxygenation (rStO2) in percent | 3 hours

SECONDARY OUTCOMES:
Reproducibility of measurement of peripheral regional tissue oxygenation (rStO2) in percent | 3 hours
Sensitivity to changes in peripheral regional tissue oxygenation (rStO2) in percent | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark